CLINICAL TRIAL: NCT04047095
Title: The Efficacy of Early Postoperative Enteral Immunonutrition on Immune Response and Outcomes in Low-Risk Cardiac Surgery Patients
Brief Title: The Efficacy of Early Postoperative Enteral Immunonutrition in Low-Risk Cardiac Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vilnius University (Other)
Responsible Party: Principal Investigator, Donata Ringaitiene, PhD Vilnius University Institute of Clinical Medicine Clinic of Anaesthesiology and Intensive Care, Vilnius University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 123
Record Dates: First submitted 2019-07-22; First posted 2019-08-06 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Cardiac Surgery
Keywords: Cardiac surgery; Immunonutrition Glutamine Bioelectrical impedance; Immunological status
MeSH Terms: interventions — Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Normal daily meals plus one sachet three times a day of immune nutrients for five days after the surgery.
  8 a.m. - normal meal plus one sachet immune nutrients
  1 p.m - normal meal plus one sachet immune nutrients 6 p.m. - normal meal plus one sachet immune nutrients
  Interventions: Dietary Supplement: Immunonutrients + normal daily meal
- Control (Active Comparator): Normal daily meals. 8 a.m. - normal meal
  1 p.m. - normal meal 6 p.m. - normal meal
  Interventions: Dietary Supplement: Normal daily meal

INTERVENTIONS:
Dietary Supplement: Immunonutrients + normal daily meal — "Glutamine Plus" by Fresenius Kabi (one sachet composition: glutamine 10 g, carbohydrate 10 g, β-carotene 1.7 mg, vitamin E 83 mg, vitamin C 250 mg, zinc 3.4 mg, selenium 50 μg, and fibre 1.2 g).
  Other Names: Normal daily meal (75-80 g protein)
  Arms: Intervention
Dietary Supplement: Normal daily meal — Normal daily meal (75-80 g protein)
  Arms: Control

SUMMARY:
The aim of this study is to investigate the efficacy of early postoperative enteral immunonutrition on immune response and outcomes in the low operative risk cardiac surgery population with low phase angle value measured by the bioelectrical impedance analysis.

DETAILED DESCRIPTION:
Study enrolls a low operative risk cardiac surgery patients who undergo elective cardiac surgery with cardiopulmonary bypass (CPB). Patient is offered to take part in a study a day prior to surgery. Information is provided regarding protocol, aim and course of study. Only signing the consent form patients could be enrolled to the study.

Study consists of:

Primary assessment - information about study. Consent form. Assessment of patient according to predefined criteria. Phase angle evaluation by bioelectrical impedance. (Day prior to surgery). It is a specific cohort of patients basically governed by surgery risk and the status of patients' cells. Euroscore II value was used to evaluate the risk of surgery. Bioelectrical impedance analysis derived phase angle was used to evaluate patients' cells frailty and vitality.

First phase of blood sampling - blood samples were taken for evaluation immunological status (cellular and humoral) and inflammatory response (CRB, complete blood count) at the surgery day morning prior to surgery.

Surgery - evaluating the course of the surgery (see exclusion criteria). Randomization - the patients will randomly selected into intervention and control groups. The patients, physicians and investigators were separate from this process. The selection sequence was computer-generated and provided to the researchers by the statistician.

Intervention - patients in the intervention group received normal daily meals plus one sachet three times a day of immune nutrients ("Glutamine Plus" by Fresenius Kabi) for five days after the surgery. The control group was provided with normal daily meals. The patients were excluded from the study if they failed to intake all of the prescribed immunonutrients.

Second phase of blood sampling - repeated taking of blood samples for evaluation immunological status (cellular and humoral) and inflammatory response (CRB, complete blood count) at the sixth day morning after the surgery.

Data collection - data is recorded (demographic data of patients, co-morbidities, instrumental parameters, phase angle values, surgery course details, immunological assesment and laboratory tests, short term and long term outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Elective cardiac surgery with cardiopulmonary bypass:
* coronary artery bypass grafting surgery (CABG);
* aortic valve replacement;
* mitral valve replacement;
* mitral valve repair;
* tricuspid valve repair;
* combined operations (CABG and valve surgery);
* Phase angle <5.5⁰ (phase angle was evaluated one day prior to surgery using bioelectrical impedance analysis (InbodyS10 device).

Exclusion Criteria:

Preoperative:

* previous cardiac surgery;
* left ventricle ejection fraction <40%;
* use of preoperative intra-aortic balloon pump (IABP);
* critical preoperative state;
* pulmonary artery mean pressure >55 mmHg;
* diagnosis of infectious endocarditis;
* pacemaker;

Operative:

* complicated intraoperative course (unplanned intervention or low cardiac output syndrome in the operating theatre: failure to wean from cardiopulmonary bypass (CPB) or intraoperative insertion of IABP or infusion of two or more inotropic medications with a cumulative dose of 0.2 mcg/kg/min);
* surgery time >6 h;
* unplanned intervention;

Postoperative:

* disturbance of dietary rules.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
CD4+ T cell | Six days
  Blood samples were collected twice on the surgery and on the sixth postoperative day by sampling blood for CD4+ T cells.
CD8+ T cell | Six days
  Blood samples were collected twice on the surgery and on the sixth postoperative day by sampling blood for CD8+ T cells.
CD69+ T cell | Six days
  Blood samples were collected twice on the surgery and on the sixth postoperative day by sampling blood for CD69+ T cells.
Interleukin-1 (IL-1) | Six days
  Blood samples were collected twice on the surgery and on the sixth postoperative day by sampling blood for IL-1.
Interleukin-6 (IL-6) | Six days
  Blood samples were collected twice on the surgery and on the sixth postoperative day by sampling blood for IL-6.
Tumor necrosis factor alfa (TNFα) | Six days
  Blood samples were collected twice on the surgery and on the sixth postoperative day by sampling blood for TNFα.

SECONDARY OUTCOMES:
Acute kidney injury | 28 days
  Short-term postoperative outcome.
Stroke | 28 days
  Short-term postoperative outcome.
ICU infectious complications | 28 days
  Short-term postoperative outcome. It was examined deep wound infections, ventilator associated and hospital acquired pneumonia, urinary tract infections, bloodstream infections, catheter-related bloodstream infections.
Duration of mechanical ventilation | 28 days
  Short-term postoperative outcome.
Retoracotomy rate | 28 days
  Short-term postoperative outcome.
Mortality | 2 years
  Long-term postoperative outcome.
Duration of hospital stay | 28 days
  Short-term postoperative outcome.
Rate of rehospitalization | 2 years
  Long-term postoperative outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jurate Sipylaite, MD, PhD, Study Chair — Vilnius University, Faculty of Medicine
Locations (1):
- Vilnius University Hospital Santaros klinikos, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Svetikiene M, Ringaitiene D, Vezeliene J, Isajevas V, Trybe D, Vicka V, Malickaite R, Jurgauskiene L, Norkuniene J, Serpytis M, Sipylaite J. The efficacy of early postoperative enteral immunonutrition on T-lymphocyte count: A randomised control study in low-risk cardiac surgery patients. Clin Nutr. 2021 Feb;40(2):372-379. doi: 10.1016/j.clnu.2020.05.009. Epub 2020 May 15. PMID 32513480